CLINICAL TRIAL: NCT05045703
Title: Characterization of Night Vision Impairment in Choroideremia and Short-Term Vitamin A Supplementation: The Dark-Adapted Retinal Function Response in Choroideremia (DARC) Study
Brief Title: The Dark-Adapted Retinal Function Response in Choroideremia (DARC) Study
Acronym: DARC
Status: Withdrawn | Phase: Not Applicable | Type: Interventional
Why Stopped: PI left the institution
Sponsor: Duke University (Other)
Collaborators: Foundation Fighting Blindness (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: Pro00108901
Record Dates: First submitted 2021-09-07; First posted 2021-09-16 (Actual); Last update posted 2023-06-29 (Actual); Status verified 2023-06

CONDITIONS: Choroideremia
Keywords: vitamin A; night vision
MeSH Terms: conditions — Choroideremia | interventions — retinol palmitate

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Vitamin A palmitate (Experimental): Vitamin A palmitate, 15,000 IU daily for 4 months
  Interventions: Dietary Supplement: Vitamin A palmitate

INTERVENTIONS:
Dietary Supplement: Vitamin A palmitate — Vitamin A palmitate, 15,000 IU daily for 4 months

SUMMARY:
Choroideremia (CHM) is an inherited retinal disorder that causes progressive vision loss, ultimately leading to complete blindness. The first symptom is generally night blindness, although, to date, little is known about the extent, type, pattern, and progression of dark-adapted visual function measures in CHM patients. We hypothesize that one of the key events causing night blindness in CHM is deficiency in the chromophore of the rod visual pigment, rhodopsin. We propose that this deficiency is at least in part due to inadequate delivery of vitamin A (all-trans-retinol) to the photoreceptors (PRs) from the ailing retinal pigment epithelium (RPE), characteristic of CHM. We hypothesize that increased availability of vitamin A would potentiate its entry into the RPE-mediated visual cycle, ultimately enabling delivery to the PRs. This would in turn allow rods to perform better by partially overcoming the RPE damage and the impaired chromophore recycling that we postulate exists in CHM. The goals of this proposal are: (1) to test the hypothesis that oral vitamin A supplementation can improve night time and peripheral vision in CHM patients, and (2) to provide detailed characterization of dark-adapted visual function outcome measures to guide interventional CHM trials.

ELIGIBILITY:
Inclusion Criteria:

* males at least 15 years of age with molecularly-confirmed diagnosis of choroideremia

Exclusion Criteria:

* inability to participate in visual field testing reliably and reproducibly

Min Age: 15 Years | Sex: Male | Healthy Volunteers: Yes
Age Groups: Child, Adult, Older Adult
Gender Based: Yes — Choroideremia is an X-linked condition that affects males almost exclusively.
Enrollment: 0 (Actual)
Dates: Start 2023-05 (Estimated); Primary Completion 2024-03 (Estimated); Study Completion 2024-05 (Estimated)

PRIMARY OUTCOMES:
Change in dark-adapted full-field visual field sensitivity | Measurements at 0, 4, and 8 months. The 0 months measurement will serve as the baseline. The 4 month measurement will assess change due to vitamin A supplementation. The 8 month measurement will assess reversal of this change following washout period
  Dark-adapted full-field visual field sensitivity will be measured using the Medmont dark-adapted chromatic perimeter.
Change in dark-adapted macular visual field sensitivity | Measurements at 0, 4, and 8 months. The 0 months measurement will serve as the baseline. The 4 month measurement will assess change due to vitamin A supplementation. The 8 month measurement will assess reversal of this change following washout period
  Dark-adapted macular visual field sensitivity will be measured using the Medmont dark-adapted chromatic perimeter.
Change in dark adaptometry | Measurements at 0, 4, and 8 months. The 0 months measurement will serve as the baseline. The 4 month measurement will assess change due to vitamin A supplementation. The 8 month measurement will assess reversal of this change following washout period
  Dark adaptometry will be measured using the MacuLogix AdaptDx dark adaptometer.

SECONDARY OUTCOMES:
Change in best corrected visual acuity | Measurements at 0, 4, and 8 months. The 0 months measurement will serve as the baseline. The 4 month measurement will assess change due to vitamin A supplementation. The 8 month measurement will assess reversal of this change following washout period
  Best corrected visual acuity will be measured using the ETDRS chart
Change in low luminance visual acuity | Measurements at 0, 4, and 8 months. The 0 months measurement will serve as the baseline. The 4 month measurement will assess change due to vitamin A supplementation. The 8 month measurement will assess reversal of this change following washout period
  Low luminance visual acuity will be measured using the ETDRS chart in low luminance conditions
Change in full-field light-adapted visual field sensitivity | Measurements at 0, 4, and 8 months. The 0 months measurement will serve as the baseline. The 4 month measurement will assess change due to vitamin A supplementation. The 8 month measurement will assess reversal of this change following washout period
  Light-adapted full-field visual field sensitivity will be measured using the Octopus 172-point GATE full-field semi-automated kinetic perimetry (SKP)
Change in light-adapted macular visual field sensitivity | Measurements at 0, 4, and 8 months. The 0 months measurement will serve as the baseline. The 4 month measurement will assess change due to vitamin A supplementation. The 8 month measurement will assess reversal of this change following washout period
  Light-adapted macular visual field sensitivity will be measured using the Centervue MAIA confocal macular microperimeter
Change in retinal pigmented epithelium (RPE) atrophy by optical coherence tomography | Measurements at 0, 4, and 8 months. The 0 months measurement will serve as the baseline. The 4 month measurement will assess change due to vitamin A supplementation. The 8 month measurement will assess reversal of this change following washout period
  Retinal pigmented epithelium (RPE) atrophy will be measured using the Spectralis macular spectral domain optical coherence tomography (SD-OCT) with and without enhanced depth imaging (EDI)
Change in retinal pigmented epithelium (RPE) atrophy by color photography | Measurements at 0, 4, and 8 months. The 0 months measurement will serve as the baseline. The 4 month measurement will assess change due to vitamin A supplementation. The 8 month measurement will assess reversal of this change following washout period
  Retinal pigmented epithelium (RPE) atrophy will be measured using the Optos wide-field color fundus photography (WF-CFP)
Change in retinal pigmented epithelium (RPE) atrophy by fundus autofluorescence | Measurements at 0, 4, and 8 months. The 0 months measurement will serve as the baseline. The 4 month measurement will assess change due to vitamin A supplementation. The 8 month measurement will assess reversal of this change following washout period
  Retinal pigmented epithelium (RPE) atrophy will be measured using the Optos wide-field fundus auto-fluorescence (WF-FAF)
Change in retinal pigmented epithelium (RPE) atrophy by fundoscopy | Measurements at 0, 4, and 8 months. The 0 months measurement will serve as the baseline. The 4 month measurement will assess change due to vitamin A supplementation. The 8 month measurement will assess reversal of this change following washout period
  Retinal pigmented epithelium (RPE) atrophy will be assessed by slit lamp biomicroscopy
Change in liver function | Measurements at 0, 4, and 8 months
  Liver function profile will be measured by laboratory using participant serum samples
Change in serum vitamin A levels | Measurements at 0, 4, and 8 months. The 0 months measurement will serve as the baseline. The 4 month measurement will assess change due to vitamin A supplementation. The 8 month measurement will assess reversal of this change following washout period
  Serum vitamin A levels will be measured by laboratory using participant serum samples

CONTACTS AND LOCATIONS:
Locations (1):
- Duke Eye Center, Durham, North Carolina, United States

IPD SHARING:
Plan to Share IPD: No